CLINICAL TRIAL: NCT03913871
Title: Text Message Program to Improve Eating Behaviors Among African Americans in New Orleans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Responsible Party: Principal Investigator, Jylana L. Sheats, Assistant Professor, Tulane University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-044-CTU
Record Dates: First submitted 2018-08-16; First posted 2019-04-12 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Diet Habit; Health Behavior; Health Knowledge, Attitudes, Practice
Keywords: mHealth; African American; Women's Health; Minority Health
MeSH Terms: conditions — Feeding Behavior; Health Behavior; Behavior

STUDY DESIGN:
Intervention Model Description: This was a clinical trial (behavioral with no clinical assessments) in which two groups of participants receive different interventions. One group received a healthy eating program, and the other group received a physical activity program.
Who Masked: Participant
Masking Description: An online randomizer software was used to assign participants into one of two arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telephone (text messages) support for healthy eating (Experimental): Participants will receive average of 1-2 text messages per day for 4 weeks focused on health eating with the aim increasing consumption of fruits, vegetables and water; and a reduce intake of sugar sweetened beverages.
  Interventions: Behavioral: Texts to support healthy eating
- Telephone (text messages) support for physical activity (Active Comparator): Participants will receive an average of 1-2 text messages per day for 4 weeks that offer physical activity and general health/wellbeing advice.
  Interventions: Behavioral: Texts to support physical activity

INTERVENTIONS:
Behavioral: Texts to support healthy eating — The intervention arm will receive tailored text messages to encourage healthy eating (increase consumption, fruits, vegetables and water; and a reduce intake of sugar sweetened beverages). Participants will receive an average of 1-2 messages per day for 4 weeks.
  Arms: Telephone (text messages) support for healthy eating
Behavioral: Texts to support physical activity — The intervention arm will receive tailored text messages to support increased minutes of physical activity per day. Participants will receive an average of 1-2 messages per day for 4 weeks.
  Arms: Telephone (text messages) support for physical activity

SUMMARY:
The purpose of this pilot study is to test the feasibility and effectiveness of a mobile phone-based text messaging intervention to change the attitudes and eating behaviors of African American women residing in New Orleans, LA.

DETAILED DESCRIPTION:
Design: The proposed study is a pre/post-test design where up to 60 female adult black/African Americans in Orleans and Jefferson Parish, Louisiana will be recruited to participated (Intervention, n=30; control n=30). If a woman is interested in participating, she will be asked to complete an evaluation/screen to determine if they are eligible for the study and asked to consent to participate. If a woman consents to participate they will be randomized to one of 2 groups:

1. Intervention group: Text messages to promote healthy eating: In this group, participants will receive personalized text messages to encourage healthy eating, specifically to increase consumption of fruits, vegetables and water; and a reduction in sugar sweetened beverages. They will receive some messages that will ask for a reply. They will receive an average of 1-2 messages per day for 4 weeks.
2. Control group: Control group participants will receive non-nutrition-related physical activity and general health/wellbeing text message. They will receive the text messages an average of 1-2 messages per day for 4 weeks

All participants will be asked to do the following tests that are not used to determine eligibility: Complete questionnaires about their background, nutrition habits, physical activity habits, health history, beliefs and opinions about health and habits. Data will be analyzed by comparing assessment outcomes within and across study arms (i.e., intervention, control).

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 25 years of age or older
2. Gender: Women
3. Ethnic background: African American or Black
4. Location: Orleans and Jefferson Parish, Louisiana
5. Own a mobile phone
6. Open to being assigned to either the intervention or control group.
7. Willing and able to use their phone to read, receive and send text messages and phone calls.
8. No overt cardiovascular disease or acute symptomatology. (self-reported).

Exclusion Criteria:

1. Age range: under 25 years of age
2. Ethnic background: not African American or Black
3. Location: Live outside of Orleans and Jefferson Parish, Louisiana
4. Does not own a mobile phone
5. Not open to being assigned to either the intervention or control group.
6. Unwilling and unable to use their phone to read, receive and send text messages and phone calls.
7. Overt cardiovascular disease or acute symptomatology. (self-reported).

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility based on self-representation of gender identity.
Enrollment: 44 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-01-11 (Actual)

PRIMARY OUTCOMES:
Fruit and vegetable intake | Baseline and 4 weeks
  Change in fruit and vegetable intake from baseline to 4 weeks as measured by self-report via the NCI Fruit and Vegetable Intake Screener (from the Eating at America's Table Study). Scale Range: Frequency of intake (fruit, vegetable) - Never (minimum) to 5+ times per day (maximum); and Portion of fruit or vegetable (cup equivalents based on dietary guidelines). To score, 1) express each reported frequency as a daily average by standardizing the midpoint of each frequency category to the number of times per day; 2) assign fruit and vegetable servings from dietary guidelines to each portion size category; and 3) compute the average daily fruit and vegetable servings for each food group by multiplying the average daily frequency (from #1) by the number of servings for the portion size (as determined in #2). To estimate the total daily number of servings, sum across all food groups (i.e., fruit and vegetable subgroups).
Beverage intake | Baseline and 4 weeks
  Change in beverage intake intake from baseline to 4 weeks as measured by self-report via the (Beverage Intake Questionnaire-15 (BEVQ-15). Scale Range: Frequency of intake (of beverage option) - Never (minimum) to 3+ times per day (maximum); Consumption (of each beverage option)- Less than 6 fl. oz. (minimum) to more than 20 fl. oz (maximum). To score the instrument, frequency ("How often") is converted to the unit of times per day, then multiplied by the amount consumed ("How much each time") to provide average daily beverage consumption in fl oz. To quantify total SSB consumption, beverage categories containing added sugars were summed (sweetened juice beverages/drinks, regular soft drinks, sweet tea, sweetened coffee, energy drinks, mixed alcoholic drinks, meal replacement beverages).

SECONDARY OUTCOMES:
Self-efficacy to improve fruit and vegetable intake | Baseline and 4 weeks
  Self-efficacy for eating fruit and vegetables as measured by self report via the Self-efficacy for fruit and vegetable survey titled Fruits and Vegetables: Pros and Cons (Norman et al., 2010). The 6-item scale is scored from Not Important (minimum) to Extremely Important (maximum). Higher scores (summed) on this scale indicated higher frequency of using change strategies for healthy eating.

CONTACTS AND LOCATIONS:
Locations (1):
- Jylana L. Sheats, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No